CLINICAL TRIAL: NCT06746558
Title: Clinical Evaluation of the Combined Effect of a Potassium Nitrate Gel and Diode Laser in the Treatment of Dentinal Hypersensitivity: a Randomized Clinical Trial
Brief Title: Potassium Nitrate Gel and Diode Laser for Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: University of Pavia (Other); University of Genova (Other)
Responsible Party: Principal Investigator, Alessandro Bruni, DDS, Orthod Spec, PhD, Research Fellow, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 76 2022-0316
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hypersensitivity Dentin
Keywords: Dentinal hypersensitivity; potassium nitrate; diode laser therapy; desensitization; dental pain management
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Potassium Nitrate Gel with Diode Laser Therapy (Experimental)
  Interventions: Combination Product: Potassium Nitrate Gel and Diode Laser Therapy
- Potassium Nitrate Gel Alone (Active Comparator)
  Interventions: Drug: Potassium Nitrate Gel Alone

INTERVENTIONS:
Combination Product: Potassium Nitrate Gel and Diode Laser Therapy — Participants in the experimental group receive treatment combining a desensitizing gel containing 5% potassium nitrate (Emoform Actisens) applied to affected teeth and diode laser therapy (980 nm). The laser is used with specific power settings (0.3W, 0.5W, 0.7W) for 20 seconds at each setting, followed by a second application of the gel and irradiation. The treatment aims to reduce dentinal hypersensitivity by occluding dentinal tubules and altering neural responses.
  Arms: Potassium Nitrate Gel with Diode Laser Therapy
Drug: Potassium Nitrate Gel Alone — Participants in the control group receive treatment with a desensitizing gel containing 5% potassium nitrate (Emoform Actisens) applied to the teeth. The gel is applied twice using a microbrush in a rubbing motion for 2 minutes each time. No diode laser therapy is administered. This intervention aims to evaluate the standalone efficacy of the gel in reducing dentinal hypersensitivity.
  Arms: Potassium Nitrate Gel Alone

SUMMARY:
The goal of this randomized clinical trial is to evaluate whether combining a potassium nitrate gel with diode laser therapy is more effective in treating dentinal hypersensitivity compared to using the gel alone. The study involves adult participants with at least two teeth affected by dentinal hypersensitivity. The main questions it aims to answer are:

Does the combined use of potassium nitrate gel and diode laser therapy reduce dentinal hypersensitivity more effectively than gel alone? How does this combined treatment impact sensitivity-related quality of life over time? Researchers will compare the outcomes between the two groups (combined therapy versus gel alone) to determine the effectiveness of the combined treatment.

Participants will:

Undergo assessments of dentinal hypersensitivity using the Shiff Air Index (SAI) and Visual Analog Scale (VAS) at baseline and at follow-ups (1 month, 3 months, and 6 months post-treatment).

Complete a questionnaire to evaluate the impact of dentinal hypersensitivity on daily life at baseline and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* At least two teeth affected by dentinal hypersensitivity.
* Good standard of home oral hygiene.

Exclusion Criteria:

* Use of pain relievers.
* Ongoing orthodontic treatment.
* Non-vital teeth or teeth with restorative materials.
* Pregnant or breastfeeding women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Reduction in Dentinal Hypersensitivity (Shiff Air Index) | Baseline (T0), immediately post-treatment (T1), 1 month (T2), 3 months (T3), and 6 months (T4)
  The Shiff Air Index measures sensitivity by applying a standardized air stimulus to the dental surface. Patients report their sensitivity level on a scale from 0 to 3, where 0 indicates no sensitivity and 3 indicates severe sensitivity. The scores are interpreted to assess the degree of dentinal hypersensitivity.
Reduction in Dentinal Hypersensitivity (Visual Analog Scale) | Baseline (T0), immediately post-treatment (T1), 1 month (T2), 3 months (T3), and 6 months (T4).
  The Visual Analog Scale (VAS) measures the intensity of pain by asking participants to rate their pain on a 10-point scale, where 0 represents no pain and 10 represents the worst pain imaginable. Participants will receive guidance to mark their pain level on the scale based on their subjective experience, providing a standardized measure of dentinal hypersensitivity.

SECONDARY OUTCOMES:
Changes in Quality of Life (Dentine Hypersensitivity Experience Questionnaire) | Baseline (T0) and 6 months (T4)
  The Dentine Hypersensitivity Experience Questionnaire (DHEQ) is a validated tool designed to assess the impact of dentinal hypersensitivity on daily activities, emotions, and overall quality of life. It consists of 15 questions rated on a 1 to 7 scale, where higher scores indicate a greater negative impact on quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Pavia, Department of Orthodontics, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simoes TM, Melo KC, Fernandes-Neto JA, Batista AL, da Silva MG, Ferreira AC, de Sousa JA, Catao MV. Use of high- and low-intensity lasers in the treatment of dentin hypersensitivity: A literature review. J Clin Exp Dent. 2021 Apr 1;13(4):e412-e417. doi: 10.4317/jced.57783. eCollection 2021 Apr. PMID 33841742
- See also: Related Info — https://portale.unipv.it/it